CLINICAL TRIAL: NCT01766687
Title: A Randomized Controlled Trial of Increased Water Intake in Chronic Kidney Disease
Brief Title: Impact of Increased Water Intake in Chronic Kidney Disease
Acronym: WIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, William Clark, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-London RCT
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; estimated glomerular filtration rate; water intake; fluid intake; renal decline
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research staff and participants were aware of the randomized group assignment; however, outcome assessors (technicians performing the laboratory measurements for the primary and secondary outcomes) are blinded to the random allocation, and the trial statistician will be blinded to patient allocation for the primary analysis
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydration (Experimental): Participants randomized to the hydration-intervention group will be asked to drink 1.0 to 1.5 L of water per day (depending on sex and weight), in addition to usual consumed beverages, for 12 months.
  Interventions: Dietary Supplement: Hydration
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Hydration
  Arms: Hydration

SUMMARY:
The investigators have designed a randomized controlled trial to test whether increased water intake slows renal decline in patients with Stage-III Chronic Kidney Disease. Participants randomized to the hydration-intervention group will be asked to drink 1.0 to 1.5 L of water per day (depending on sex and weight), in addition to usual fluid intake, for one year. The investigators will calculate the change in kidney function (estimated glomerular filtration rate, measured every three months for 12 months), and compare renal decline between the intervention and control groups. The investigators hypothesize that increased water intake will slow renal decline.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Able to provide informed consent and willing to complete follow-up visits.
* Estimated glomerular filtration rate between 30 and 60 ml/min/1.73m2
* Trace protein or greater (Albustix) or urine albumin/creatinine ratio >2.8 mg/mmol (if female) or >2.0 mg/mmol (if male) from a random spot urine sample

Exclusion Criteria:

* Self-reported fluid intake >10 cups/day or 24-hr urine volume >3L.
* Enrolled in another trial that could influence the intervention, outcomes or data collection of this trial (or previously enrolled in this trial)
* Received one or more dialysis treatments in the past month
* Kidney transplant within past six months (or on waiting list)
* Pregnant or breastfeeding
* History of kidney stones in past 5 years
* Less than two years life expectancy
* Serum sodium <130 mEq/L without suitable explanation
* Serum calcium >2.6 mmol/L without suitable explanation
* Currently taking hydrochlorothiazide >25 mg/d, indapamide >1.25 mg/d, furosemide >40 mg, or metolazone >2.5 mg/d
* Currently taking lithium
* Patient is under fluid restriction (<1.5 L a day) for kidney disease, heart failure, or liver disease, AND meets any of the following criteria: i) end stage of the disease (heart left ventricular ejection fraction <40%, NYHA class 3 or 4, or end stage cirrhosis) or ii) hospitalization secondary to heart failure, ascites and/or anasarca
* Patient has GI disease (history of inflammatory bowel disease, Crohns, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2013-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Renal decline | Baseline and 12 months
  Change in estimated glomerular filtration rate between baseline and 12 months

SECONDARY OUTCOMES:
24-hour urine albumin | Baseline and 12 months
  Change in 24-hour urine albumin between baseline and 12 months
Rapid renal decline | Baseline and 12 months
  Proportion with eGFR (estimated glomerular filtration rate) decline >5% between baseline and 12 months
Measured creatinine clearance | Baseline and 12 months
  Change in measured creatinine clearance between baseline and 12 months
Health-related quality of life | Baseline and 12 months
  Change in health-related quality of life between baseline and 12 months
Copeptin | Baseline and 12 months
  Change in copeptin between baseline and 12 months

OTHER OUTCOMES:
Body Mass Index | Baseline and 12 months
  Change in Body Mass Index between baseline and 12 months
Blood pressure | Baseline and 12 months
  Change in mean arterial blood pressure between baseline and 12 months
HbA1c | Baseline and 12 months
  Change in HbA1c between between baseline and 12 months
Long-term renal decline | Baseline and 24 months
  Change in estimated glomerular filtration rate between baseline and 24 months
Effect of fluid coaching on adherence | 12 and 24 months
  Change in urine volume between 12 months and 24-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: William F Clark, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Clark WF, Huang SH, Garg AX, Gallo K, House AA, Moist L, Weir MA, Sontrop JM. The Chronic Kidney Disease Water Intake Trial: Protocol of a Randomized Controlled Trial. Can J Kidney Health Dis. 2017 Aug 22;4:2054358117725106. doi: 10.1177/2054358117725106. eCollection 2017. PMID 28856009
- [Derived] Moist LM. Can Additional Water a Day Keep the Cysts Away, in Patients with Polycystic Kidney Disease? NEJM Evid. 2022 Jan;1(1):EVIDe2100027. doi: 10.1056/EVIDe2100027. Epub 2021 Nov 4. PMID 38320097
- [Derived] Clark WF, Sontrop JM, Huang SH, Gallo K, Moist L, House AA, Cuerden MS, Weir MA, Bagga A, Brimble S, Burke A, Muirhead N, Pandeya S, Garg AX. Effect of Coaching to Increase Water Intake on Kidney Function Decline in Adults With Chronic Kidney Disease: The CKD WIT Randomized Clinical Trial. JAMA. 2018 May 8;319(18):1870-1879. doi: 10.1001/jama.2018.4930. PMID 29801012
- [Derived] Roussel R, Velho G, Bankir L. Vasopressin and diabetic nephropathy. Curr Opin Nephrol Hypertens. 2017 Jul;26(4):311-318. doi: 10.1097/MNH.0000000000000335. PMID 28403013